CLINICAL TRIAL: NCT00965744
Title: A Clinical Trial of the Vessel Sealing System (LigaSure) in Azygoportal Disconnection and Splenectomy in Patients With Portal Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Changzheng Hospital (Other)
Responsible Party: Qiang Wang, MD, Shanghai Chang Zheng Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SCZH-0908-016
Record Dates: First submitted 2009-08-25; First posted 2009-08-26 (Estimated); Last update posted 2009-08-27 (Estimated); Status verified 2009-08

CONDITIONS: Liver Cirrhosis
Keywords: Ligasure vessel sealing system; Azygoportal Disconnection; Splenectomy; Portal hypertension
MeSH Terms: conditions — Liver Cirrhosis; Hypertension, Portal

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vessel sealing system LigaSure (VS group) (Experimental): Patients in VS group undergoing esophagogastric decongestion (Azygoportal Disconnection) and splenectomy with or without esophageal transaction with the vessel sealing system LigaSure.
  Interventions: Device: Vessel sealing system LigaSure
- Conventional hand-tied method (CH group) (No Intervention): Patients in CH group undergoing esophagogastric decongestion (Azygoportal Disconnection) and splenectomy with or without esophageal transaction with the conventional hand-tied method.

INTERVENTIONS:
Device: Vessel sealing system LigaSure — Patients in VS group undergoing esophagogastric decongestion (Azygoportal Disconnection) and splenectomy with or without esophageal transaction with the vessel sealing system LigaSure.
  Arms: Vessel sealing system LigaSure (VS group)

SUMMARY:
The aim of this trial was to verify the efficiency of a new surgical device (the LigaSure vessels sealing system) in esophagogastric decongestion and splenectomy in patients with portal hypertension.

DETAILED DESCRIPTION:
Bleeding from esophageal and gastric cardia varices is the major life threatening complication in patients with portal hypertension. Patients with portal hypertension have a mortality rate of 30%-50% at the first episode of esophagogastric variceal rupture. The associated 1-year mortality rate is reported to be 75%. The ideal treatment for gastric varices should effectively control bleeding and improve the liver function to optimum levels. Although endoscopic treatments have showed great promise for esophageal varices, there is still controversy regarding the treatment of gastric varices. Hepatic encephalopathy remain a dominant problems after transjugular intrahepatic portosystemic shunt placement (TIPS) and surgical shunts. A meta-analysis has shown that the incidence of hepatic encephalopathy and mortality was increased significantly either in nonselective or selective shunt operations.

Esophagogastric decongestion and splenectomy with or without esophageal transaction were the fundamental operation performed in our department for patients with portal hypertension. Patients under the azygoportal devascularization methods revealed reduction of the encephalopathy as well as diminished rebleeding rates. The crucial point of the procedure is prevention of the brisk bleeding from the dilated vessels like enlarged azygoportal collaterals. Conventional hand-tied ligatures can become dislodged and represent a foreign body, and more important, it is tedious and time-consuming. The LigaSure vessel sealing system (Valleylab, Boulder, Colorado) is a bipolar electrosurgical device, sealing vessels up to 7 mm in diameter, by denaturing collagen and elastin within vessel wall and surrounding connective tissue. This device was tested, with excellent results, in different fields of surgery (gastrointestinal, hepatopancreatobiliary, urologic, gynecologic, laparoscopic, etc), as demonstrated by several recently published studies. Shamiyeh et al confirmed the reliability of LigaSure for the closure of the veins in laparoscopic azygoportal disconnection procedure on the portal hypertension porcine model in 2005, there was no intra- or post-operative bleeding and no conversion to open surgery, and when more than 2 mm far from the thermal energy source, no collateral damage of the solid tissue such as stomach could be detected.

ELIGIBILITY:
Inclusion Criteria:

* Patients with liver cirrhosis accompanied by portal hypertension and secondary hypersplenism due to hepatitis, alcoholic cirrhosis or schistosomiasis, who undergoing elective azygoportal disconnection and splenectomy

Exclusion Criteria:

* Liver function as Child-Pugh C
* Hemoglobin < 9 g/dL
* Ascites
* Abnormal coagulation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2006-01; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Operating time, from the skin incision to the final skin closure. Intraoperative blood loss, calculated by a graduated suction device and by amounts of blood involved into the sponges by the end of the operation. | Within the operation

SECONDARY OUTCOMES:
Postoperative drainage volume, complications (spleen fever, bleeding and portal vein thrombosis), length of incision, postoperative pain and time to discharge. | within the first 30 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Qiang Wang, MD, Study Chair — Shanghai Chang Zheng Hospital; Jia Dong Gao, MD, Principal Investigator — Department of General Surgery, Shanghai Chang Zheng Hospital; Wei Jun Wang, MD, Principal Investigator — Department of General Surgery, Shanghai Chang Zheng Hospital; Hou Shan Yao, MD, Principal Investigator — Department of General Surgery, Shanghai Chang Zheng Hospital; Zhi Qian Hu, MD, Principal Investigator — Department of General Surgery, Shanghai Chang Zheng Hospital
Locations (1):
- Department of General Surgery, Shanghai Chang Zheng Hospital, Shanghai, Shanghai Municipality, China